CLINICAL TRIAL: NCT00022087
Title: Phase III Trial of Intravenous Zoledronic Acid (Zometa) in the Prevention of Bone Loss in Localized Breast Cancer Patients With Chemotherapy-Induced Ovarian Failure
Brief Title: Zoledronate, Calcium, and Vitamin D in Preventing Bone Loss in Women Receiving Adjuvant Chemotherapy for Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CALGB-79809; U10CA031946 (NIH); CALGB-79809; NCI-P01-0184; CDR0000068781 (Registry Identifier: NCI Physicians Data Query)
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: osteoporosis; stage I breast cancer; stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis | interventions — Cholecalciferol; Vitamin D; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoledronic acid initial tx (Experimental): Zoledronic acid + calcium + Vit D for 2 years, followed by Calcium + vit D for 1 year
  Interventions: Dietary Supplement: calcium salts; Dietary Supplement: cholecalciferol; Drug: zoledronic acid
- Calcium + Vit D initial Tx (Experimental): Calcium + vitamin D for 1 year followed by zoledronic acid + calcium + vit D for 2 years
  Interventions: Dietary Supplement: calcium salts; Dietary Supplement: cholecalciferol; Drug: zoledronic acid

INTERVENTIONS:
Dietary Supplement: calcium salts — 1000 mg PO per day
Dietary Supplement: cholecalciferol — 400 IU PO per day
  Other Names: Vitamin D
Drug: zoledronic acid — 4 mg IV infusion q 3 months, months 1-24 in Zoledronic acid initial tx arm and months 13-36 in calcium + vit D initial tx arm
  Other Names: Zometa

SUMMARY:
RATIONALE: Zoledronate plus calcium and vitamin D may prevent bone loss in patients receiving adjuvant chemotherapy for breast cancer. It is not yet known which regimen is more effective in preventing bone loss.

PURPOSE: This randomized phase III trial is comparing two regimens of zoledronate plus calcium and vitamin D to see how well they work in preventing bone loss in women who are receiving adjuvant chemotherapy for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the bone mineral density in the lumbar spine after 12 and 36 months of therapy with zoledronate, calcium, and cholecalciferol (vitamin D) in women with breast cancer receiving adjuvant chemotherapy.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to intent to treat with tamoxifen (yes vs no) and node status (negative vs positive vs unknown [for patients receiving neoadjuvant therapy]). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Beginning on the first day of adjuvant chemotherapy (or within 3 months after the first day), patients receive zoledronate IV over at least 15 minutes once every 3 months during months 1-24 and oral calcium and oral cholecalciferol (vitamin D) daily during months 1-36.
* Arm II: Beginning on the first day of adjuvant chemotherapy (or within 3 months after the first day), patients receive oral calcium and oral vitamin D daily during months 1-36 and zoledronate IV over at least 15 minutes once every 3 months during months 13-36.

PROJECTED ACCRUAL: Approximately 400 patients (200 per treatment arm) will be accrued for this study within 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast by fine needle aspirate, biopsy (tru-cut, core, stereotactic), lumpectomy, or modified radical mastectomy

  * Stage I-III (any T, any N, M0)
  * Stage IV due solely to supraclavicular node involvement allowed
* Plan to use adjuvant chemotherapy* with or without adjuvant endocrine therapy*

  * Subsequent adjuvant hormonal therapy with an aromatase inhibitor allowed in women rendered postmenopausal by adjuvant chemotherapy NOTE: *Must be specified prior to study entry
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 40 and over

Sex:

* Female

Menopausal status:

* See Disease Characteristics
* Premenopausal, defined as actively menstruating or last menstrual period occurred within 6 months prior to study entry

  * Prior hysterectomy without bilateral oophorectomy and estradiol and follicle-stimulating hormone within premenopausal range prior to the initiation of chemotherapy allowed

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No more than 3 months since prior adjuvant chemotherapy

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics
* See Menopausal status

Other:

* No other concurrent bisphosphonates
* No concurrent digoxin
* No concurrent tetracycline
* Concurrent neoadjuvant therapy allowed
* Concurrent enrollment on therapeutic adjuvant clinical trials allowed provided the therapeutic trial does not preclude participation in this trial

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2001-12; Primary Completion 2007-03 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Bone mineral density in the lumbar spine | 12 months from randomization

SECONDARY OUTCOMES:
Bone mineral density in the lumbar spine | 36 months post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Shapiro, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (107):
- United States (107):
  - Arroyo Grande Community Hospital, Arroyo Grande, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - El Camino Hospital, Mountain View, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - Kent General Hospital at Bayhealth Medical Center, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - St. Francis Hospital, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Cancer Research Network, Incorporated, Plantation, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Suniti Medical Corporation, Merrillville, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Central Maine Medical Center, Lewiston, Maine
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Union Hospital Cancer Center at Union Hospital, Elkton MD, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts
  - Bethke Cancer Center at Emerson Hospital, Concord, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Saint Luke's Hospital, Chesterfield, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Missouri Cancer Care, P. C. - Wentzville, Wentzville, Missouri
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Oncology Center at St. Joseph Hospital, Nashua, New Hampshire
  - Jersey City Medical Center at Liberty Health, Jersey City, New Jersey
  - Cancer Institute of New Jersey at the Cooper University Hospital - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - Community General Hospital of Greater Syracuse, Syracuse, New York
  - Faxton Regional Cancer Center, Utica, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Miriam Hospital at Lifespan, Providence, Rhode Island
  - CCOP - Greenville, Greenville, South Carolina
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Community Cancer Center at Rutland Regional Medical Center, Rutland, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - St. Mary's Regional Cancer Center at St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- [Result] Shapiro CL, Halabi S, Gibson G, et al.: Effect of zoledronic acid (ZA) on bone mineral density (BMD) in premenopausal women who develop ovarian failure (OF) due to adjuvant chemotherapy (AdC): first results from CALGB trial 79809. [Abstract] J Clin Oncol 26 (Suppl 15): A-512, 2008.
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716